CLINICAL TRIAL: NCT02520596
Title: Bioavailability of Anthocyanins in Humans Following the Ingestion of Berries and Grapes
Brief Title: Absorption and Metabolism of Dietary Phenolics From Raspberries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Collaborators: University of Glasgow (Other); National Processed Raspberry Council (Unknown)
Responsible Party: Principal Investigator, Daniele Del Rio, Associate Professor, University of Parma
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DDR-002
Record Dates: First submitted 2015-07-31; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Dietary Modifications
Keywords: Raspberries; Anthocyanins; Ellagitannins; Metabolites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Bioavailability of Raspberry polyphenols

SUMMARY:
Red raspberries are a rich source of (poly)phenolic compounds, the main components being anthocyanins and ellagitannins. There is growing evidence linking consumption of these compounds with beneficial effects on human health. However, the mechanisms involved remain poorly understood principally because of a limited understanding of the bioavailability of ellagitannins and anthocyanins. This study aims to explore the identity and amounts of the phenolic metabolites of anthocyanins and ellagitannins in human plasma and urine following acute ingestion of raspberries. For this purpose ten healthy volunteers were feed 300 g of blended raspberries containing in total 293 μmol anthocyanins and 250 μmol ellagitannins. All urine excreted over 48 h after the ingestion of raspberries was collected and blood samples were collected before (0 h) and after raspberry consumption up to 24 h. Metabolites were identified and quantified by ultra high performance liquid chromatography-mass spectrometry (UHPLC-MS).

ELIGIBILITY:
Inclusion Criteria:

* in general good health

Exclusion Criteria:

* smoking
* pregnancy
* vegetarian
* sustained use of nutritional supplements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Changes in urinary anthocyanin and ellagitannin metabolite excretion after ingestion of 300g blended raspberries measured by ultra-high performance liquid chromatography-mass spectrometry | baseline excretion (12 h before intervention), and 0-4 h, 4-8 h, 8-24 h, 24-32 h, 32-48 h post ingestion
  All urine excreted for 12 h prior to supplementation was collected as well as that excreted over 48 h after ingestion of raspberries. Urine samples were vortexed, centrifuged at 16110 g for 10 min at 5°C, and passed through 0.45 μm filter discs prior to the analysis of 5 μL aliquots by UHPLC-MS.

SECONDARY OUTCOMES:
Changes in plasma concentration of anthocyanin and ellagitannin metabolites after ingestion of 300g blended raspberries measured by ultra-high performance liquid chromatography-mass spectrometry | 0 h, 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 24 h post ingestion
  Blood samples were collected in heparin tubes before and after raspberry consumption up to 24 h. Plasma samples were vortexed and 400 µL aliquots were mixed with 1 mL of 2% formic acid in acetonitrile. The samples were then vortexed and ultrasonicated for 10 min. After centrifugation at 16110 g for 10 min, supernatants were reduced to dryness in vacuo using a Speedvac concentrator and resuspended in 100 µL of methanol:water:formic acid (50:50:0.1, v/v/v) which was centrifuged at 16100 g for 10 min and 5 μL aliquots of the supernatant analysed by UHPLC-MS.

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Del Rio, PhD, Principal Investigator — University of Parma
Locations (1):
- University of Parma - Department of Food Science, Parma, Italy

REFERENCES:
- [Background] Gonzalez-Barrio R, Borges G, Mullen W, Crozier A. Bioavailability of anthocyanins and ellagitannins following consumption of raspberries by healthy humans and subjects with an ileostomy. J Agric Food Chem. 2010 Apr 14;58(7):3933-9. doi: 10.1021/jf100315d. PMID 20218618
- [Background] Gonzalez-Barrio R, Edwards CA, Crozier A. Colonic catabolism of ellagitannins, ellagic acid, and raspberry anthocyanins: in vivo and in vitro studies. Drug Metab Dispos. 2011 Sep;39(9):1680-8. doi: 10.1124/dmd.111.039651. Epub 2011 May 27. PMID 21622625
- [Background] Stalmach A, Edwards CA, Wightman JD, Crozier A. Gastrointestinal stability and bioavailability of (poly)phenolic compounds following ingestion of Concord grape juice by humans. Mol Nutr Food Res. 2012 Mar;56(3):497-509. doi: 10.1002/mnfr.201100566. Epub 2012 Feb 14. PMID 22331633
- [Background] Fang J. Some anthocyanins could be efficiently absorbed across the gastrointestinal mucosa: extensive presystemic metabolism reduces apparent bioavailability. J Agric Food Chem. 2014 May 7;62(18):3904-11. doi: 10.1021/jf405356b. Epub 2014 Mar 31. PMID 24650097
- [Background] de Ferrars RM, Czank C, Zhang Q, Botting NP, Kroon PA, Cassidy A, Kay CD. The pharmacokinetics of anthocyanins and their metabolites in humans. Br J Pharmacol. 2014 Jul;171(13):3268-82. doi: 10.1111/bph.12676. PMID 24602005
- [Background] Czank C, Cassidy A, Zhang Q, Morrison DJ, Preston T, Kroon PA, Botting NP, Kay CD. Human metabolism and elimination of the anthocyanin, cyanidin-3-glucoside: a (13)C-tracer study. Am J Clin Nutr. 2013 May;97(5):995-1003. doi: 10.3945/ajcn.112.049247. PMID 23604435
- [Background] Cassidy A, Mukamal KJ, Liu L, Franz M, Eliassen AH, Rimm EB. High anthocyanin intake is associated with a reduced risk of myocardial infarction in young and middle-aged women. Circulation. 2013 Jan 15;127(2):188-96. doi: 10.1161/CIRCULATIONAHA.112.122408. PMID 23319811
- [Background] Del Rio D, Rodriguez-Mateos A, Spencer JP, Tognolini M, Borges G, Crozier A. Dietary (poly)phenolics in human health: structures, bioavailability, and evidence of protective effects against chronic diseases. Antioxid Redox Signal. 2013 May 10;18(14):1818-92. doi: 10.1089/ars.2012.4581. Epub 2012 Aug 27. PMID 22794138
- [Background] Stalmach A, Edwards CA, Wightman JD, Crozier A. Identification of (poly)phenolic compounds in concord grape juice and their metabolites in human plasma and urine after juice consumption. J Agric Food Chem. 2011 Sep 14;59(17):9512-22. doi: 10.1021/jf2015039. Epub 2011 Aug 12. PMID 21812481